CLINICAL TRIAL: NCT05130463
Title: A Regulatory Requirement Non-interventional Study to Monitor the Safety and Effectiveness of Esgliteo (Empagliflozin/Linagliptin, 10/5mg, 25/5mg) in Korean Patients With Type 2 Diabetes Mellitus
Brief Title: Esgliteo Post Marketing Surveillance (PMS) in Korean Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1275-0028
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Linagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with type 2 diabetes mellitus: Patients aged 19 years or older, diagnosed with type 2 diabetes mellitus in Korea, who initiated treatment with ESGLITEO® for the first time in accordance with the locally approved label.
  Interventions: Drug: Empagliflozin/Linagliptin

INTERVENTIONS:
Drug: Empagliflozin/Linagliptin — Participants received Empagliflozin 10mg or 25mg and Linagliptin 5mg (Fixed Dose) Film-coated tablets orally once daily with or without food.
  Other Names: Esgliteo®

SUMMARY:
The objectives of this study are to monitor the safety and effectiveness of Esgliteo in Korean patients with type 2 diabetes mellitus in a routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have started at first time on Esgliteo in accordance with the approved label in Korea
* Age ≥19 years at enrolment
* Patients who have signed on the data release consent form

Exclusion Criteria:

* Patients with previous exposure to Esgliteo
* Patients with hypersensitivity to the empagliflozin and/or linagliptin or any of the excipients
* Patients with type 1 diabetes or diabetic ketoacidosis
* Patients with estimated Glomerular Filtration Rate (eGFR) < 45 mL/min/1.73m2, end stage renal disease, or patient on dialysis
* Patients for whom empagliflozin/linagliptin is contraindicated according to the local label of Esgliteo

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 2 diabetes mellitus in Korea.
Sampling Method: Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- South Korea (30):
  - Cheonan Chungmu Hospital, Cheonan-si, Chungcheongnam-do
  - Woori-hospital, Bucheon-si, Gyeonggi-do
  - Seo Jung Hwa Internal medicine, Gwangmyeong, Gyeonggi-do
  - Samsung Internal medicine, Hanam, Gyeonggi-do
  - Brrunmadi Orthopedics, Seongnam-si, Gyeonggi-do
  - ST.Mary's Will Hospital, Seongnam-si, Gyeonggi-do
  - 21Chospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Dr.Yoon's Clinic, Gyeongsan-si, Gyeongsangbuk-do
  - Yeongju gidok hospital, Yeongju, Gyeongsangbuk-do
  - Seoul NIM Clinic, Changwon-si,, Gyeongsangnam-do
  - Choi Bongki Internal Medicine, Changwon-si, Gyeongsangnam-do
  - Gyeongsang National Univ. Changwon Hospital, Changwon-si, Gyeongsangnam-do
  - Chonnam National Univ. Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Park Chang Hyun Clinic, Mokpo-si, Jeollanam-do
  - Mokpo Gospel Internal Medicine Clinic, Mokpo-si, Jeollanam-do
  - Park Il Jong Clinic, Mokpo-si, Jeollanam-do
  - Yeosu Jeil Hospital, Yeosu, Jeollanam-do
  - Yonsei Clinic, Busan
  - MyungJi Medical Center, Busan
  - Choi Won Rak Clinic, Busan
  - Daejeon Endo Internal Medicine, Daejeon
  - Good Morning Interanl medicine, Gwangju
  - Park Clinic, Gwangju
  - IBS Medical Clinic, Incheon
  - Dream Internal Medicine Clinic, Jeju City
  - D&F Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Yonsei Checkup Clinic, Seoul
  - CBY Endocrine & Internal Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional, multi-centre, single-country study focuses on providing additional safety and effectiveness information for Korean patients with type 2 diabetes mellitus in routine clinical settings. It aims to monitor the safety and effectiveness of ESGLITEO® (Empagliflozin/Linagliptin, 10/5 mg, 25/5 mg) in these patients as part of post-marketing surveillance.
Pre-assignment Details: Patients diagnosed with type 2 diabetes mellitus in Korea were included in this study. ESGLITEO® is administered as an adjunct to diet and exercise therapy to improve glycaemic control in these patients. This non-interventional study (NIS) follows a single-arm design with ESGLITEO®, prescribed according to the local label and at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Patients Diagnosed With Type 2 Diabetes Mellitus
Started | 1053
Completed | 616
Not Completed | 437
Not completed — Unspecified reasons | 2
Not completed — off-label indication dose | 435

BASELINE CHARACTERISTICS:
Population: Safety Set: This set includes participants who signed the data release consent form, took Esgliteo at least once, and were followed up by a physician at least once.
Arm/Group | Patients Diagnosed With Type 2 Diabetes Mellitus
Number analyzed (Participants) | 616
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants Whose CRF Was Retrieved: This includes participants who signed the data release consent form, participated in the study, and took Esgliteo at least once.
  years | 58.7 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants Whose CRF Was Retrieved: This includes participants who signed the data release consent form, participated in the study, and took Esgliteo at least once.
  Participants
    Female | 230
    Male | 386
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants Whose CRF Was Retrieved: This includes participants who signed the data release consent form, participated in the study, and took Esgliteo at least once.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 616
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants Whose CRF Was Retrieved: This includes participants who signed the data release consent form, participated in the study, and took Esgliteo at least once.
  Participants
    American Indian or Alaska Native | 0
    Asian | 616
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Baseline glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage] — Baseline HbA1c values for participants who took Esgliteo at least once, and were evaluated for the effectiveness is presented. Population: These cases include those who signed the data release consent form to participate in this study as subject, visited as per the study schedule, took Esgliteo at least once, and were evaluated for the effectiveness.
  Percentage
    number analyzed (Participants) | 342
    (all) | 7.32 (1.191)

OUTCOME MEASURES:

1. Primary Outcome: All Reported Adverse Events Collected From Subjects Taking at Least One Dose of ESGLITEO®
Description: These include those who signed the data release consent form to participate in this study as subject, took Esgliteo once at least, and were followed up by the physician once or more.
Time Frame: From first trial drug administration up to 24 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Number of events
Groups:
- Patients Diagnosed With Type 2 Diabetes: Patients aged 19 years or older, diagnosed with type 2 diabetes mellitus in Korea, who initiated treatment with ESGLITEO® for the first time in accordance with the locally approved label.
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 616
Number of events | 26

2. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) After 12 Weeks of Treatment
Description: The mean change from baseline in glycosylated hemoglobin (HbA1c) after 12 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: Effectiveness Set: Participants who signed the data release consent form, followed the study schedule, took Esgliteo at least once, and were evaluated for effectiveness.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 303
Percentage | -0.21 (1.126)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; Test type: Other; p = 0.0011, t-test, 2 sided — Comparison of the change in HbA1c from baseline to the values at 12 weeks post Esgliteo administration

3. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) After 24 Weeks of Treatment
Description: The mean change from baseline in glycosylated hemoglobin (HbA1c) after 24 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 139
Percentage | -0.27 (0.983)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; Test type: Other; p = 0.0014, t-test, 2 sided — Comparison of the change in HbA1c from baseline to the values at 24 weeks post Esgliteo administration

4. Secondary Outcome: Percentage of Participants With HbA1c Reaching Less Than 7% From Baseline (Target Effectiveness Response Rate) After 12 Weeks of Treatment
Description: The percentage of patients whose glycosylated hemoglobin (HbA1c) levels dropped below 7% at 12 weeks following trial drug administration are presented.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 303
Percentage of participants | 49.50 [43.74 to 55.28]

5. Secondary Outcome: Percentage of Participants With HbA1c Reaching Less Than 7% From Baseline (Target Effectiveness Response Rate) After 24 Weeks of Treatment
Description: The percentage of patients whose glycosylated hemoglobin (HbA1c) levels dropped below 7% at 24 weeks following trial drug administration are presented.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 139
Percentage of participants | 53.24 [44.59 to 61.74]

6. Secondary Outcome: Percentage of Participants With Occurrence of Relative Effectiveness Response After 12 Weeks of Treatment
Description: Relative effectiveness was defined as participants whose HbA1c decreased by at least 0.5% (relative effectiveness response rate) at 12 weeks after administration of ESGLITEO®.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 303
Percentage of participants | 29.37 [24.30 to 34.85]

7. Secondary Outcome: Percentage of Participants With Occurrence of Relative Effectiveness Response After 24 Weeks of Treatment
Description: Relative effectiveness was defined as participants whose HbA1c decreased by at least 0.5% (relative effectiveness response rate) at 24 weeks after administration of ESGLITEO®.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 139
Percentage of participants | 38.85 [30.71 to 47.48]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 12 Weeks of Treatment
Description: Change from baseline in fasting plasma glucose (FPG) of participants after 12 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 302
milligrams per deciliter (mg/dL) | -10.8 (54.90)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; FPG at baseline vs FPG after 12 weeks of treatment; Test type: Other; p = 0.0008, t-test, 2 sided — Comparison of the change in FPG from baseline to the values at 12 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks of Treatment
Description: Change from baseline in fasting plasma glucose (FPG) of participants after 24 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 154
milligrams per deciliter (mg/dL) | -12.3 (55.76)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; FPG at baseline vs FPG after 24 weeks of treatment; Test type: Other; p = 0.0068, t-test, 2 sided — Comparison of the change in FPG from baseline to the values at 24 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

10. Secondary Outcome: Change From Baseline in Body Weight After 12 Weeks of Treatment
Description: Change from baseline in body weight of participants after 12 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 107
Kilogram (kg) | -0.72 (5.583)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; Body weight at baseline vs Body weight after 12 weeks of treatment; Test type: Other; p = 0.1867, t-test, 2 sided — Comparison of the change in body weight from baseline to the values at 12 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

11. Secondary Outcome: Change From Baseline in Body Weight After 24 Weeks of Treatment
Description: Change from baseline in body weight of participants after 24 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 93
Kilogram (kg) | -1.27 (3.204)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; Body weight at baseline vs Body weight after 24 weeks of treatment; Test type: Other; p = 0.0003, t-test, 2 sided — Comparison of the change in body weight from baseline to the values at 24 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

12. Secondary Outcome: Change From Baseline in Blood Pressure (Systolic Blood Pressure [SBP], Diastolic Blood Pressure [DBP]) After 12 Weeks of Treatment
Description: Mean change from baseline in blood pressure (systolic blood pressure [SBP], diastolic blood pressure [DBP]) of participants after 12 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 241
Millimeters of mercury (mmHg)
  Change from baseline in systolic blood pressure after 12 weeks of treatment | -2.8 (13.77)
  Change from baseline in diastolic blood pressure after 12 weeks of treatment | -1.6 (9.91)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; SBP at baseline vs SBP after 12 weeks of treatment; Test type: Other; p = 0.0020, t-test, 2 sided — Comparison of the change in SBP from baseline to the values at 12 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level
Statistical Analysis 2: Comparison: Patients Diagnosed With Type 2 Diabetes; DBP at baseline vs DBP after 12 weeks of treatment; Test type: Other; p = 0.0132, t-test, 2 sided — Comparison of the change in DBP from baseline to the values at 12 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

13. Secondary Outcome: Change From Baseline in Blood Pressure (Systolic Blood Pressure [SBP], Diastolic Blood Pressure [DBP]) After 24 Weeks of Treatment
Description: Mean change from baseline in blood pressure (systolic blood pressure [SBP], diastolic blood pressure [DBP]) of participants after 24 weeks of treatment is presented.
Time Frame: From the first trial drug administration up to 24 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Patients Diagnosed With Type 2 Diabetes
Number analyzed (Participants) | 134
Millimeters of mercury (mmHg)
  Change from baseline in systolic blood pressure after 24 weeks of treatment | -0.4 (16.59)
  Change from baseline in diastolic blood pressure after 24 weeks of treatment | -0.6 (11.01)
Statistical Analysis 1: Comparison: Patients Diagnosed With Type 2 Diabetes; SBP at baseline vs SBP after 24 weeks of treatment; Test type: Other; p = 0.7591, t-test, 2 sided — Comparison of the change in SBP from baseline to the values at 24 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level
Statistical Analysis 2: Comparison: Patients Diagnosed With Type 2 Diabetes; DBP at baseline vs DBP after 24 weeks of treatment; Test type: Other; p = 0.5161, t-test, 2 sided — Comparison of the change in DBP from baseline to the values at 24 weeks post Esgliteo administration; Paired t-test: Statistically significant at a 5% two-sided level

ADVERSE EVENTS:
Time Frame: AE and All-cause mortality collection period: From first Esgliteo administration up to 24 weeks.
Description: Safety Set: This set includes participants who signed the data release consent form, took Esgliteo at least once, and were followed up by a physician at least once.
Arm/Group | Patients Diagnosed With Type 2 Diabetes
All-Cause Mortality (participants affected / at risk) | 0/616
Serious Adverse Events (participants affected / at risk) | 3/616
Other Adverse Events (participants affected / at risk) | 0/616
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Diagnosed With Type 2 Diabetes (N=616)
Adrenal insufficiency (Endocrine disorders) | 1
Aortic thrombosis (Vascular disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT05130463/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT05130463/SAP_001.pdf